CLINICAL TRIAL: NCT07345325
Title: Rifampin-free Regimen Versus Rifampin-containing Regimen in the Treatment of Staphylococcal Prosthetic Valve Endocarditis: a Multicenter Randomized Controlled Non-inferiority Study
Brief Title: Rifampin-free Regimen Versus Rifampin-containing Regimen in the Treatment of Staphylococcal Prosthetic Valve Endocarditis
Acronym: RIFREE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC24_0404; 2024-518018-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Infective Endocarditis
Keywords: infective endocarditis; prosthetic valve; Rifampin; Staphylococcus aureus
MeSH Terms: conditions — Endocarditis; Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifampin-free regimen. (Experimental): The experimental arm of the study involves the removal of rifampicin from the antibiotic regimen recommended by the 2023 ESC (European Society of Cardiology) guidelines and the 2025 French guidelines (AEPEI/SPILF) for the treatment of staphylococcal prosthetic valve endocarditis.
  Interventions: Drug: Rifampin-free regimen
- Rifampin containing regimen (Active Comparator): Rifampin containing regimen (900 mg/day). Antibiotic treatment of endocarditis in accordance with the 2023 ESC guidelines and the 2025 French guidelines (AEPEI/SPILF).
  Interventions: Drug: Rifampin containing regimen

INTERVENTIONS:
Drug: Rifampin-free regimen — Rifampin-free regimen. The choice of other antibiotics is at the discretion of the physicians in charge but should be in accordance with the 2023 ESC guidelines and 2025 French guidelines (AEPEI/SPILF).
  Arms: Rifampin-free regimen.
Drug: Rifampin containing regimen — Rifampin containing regimen (900 mg/day). Antibiotic treatment of endocarditis in accordance with the 2023 ESC guidelines and 2025 French guidelines.
  Arms: Rifampin containing regimen

SUMMARY:
The primary objective of this study is to demonstrate that a rifampin-free regimen is non-inferior to the rifampin-containing regimen in terms of all-cause mortality in staphylococcal prosthetic valve endocarditis within 6 months after randomization.

DETAILED DESCRIPTION:
A rifampin-based treatment is recommended for prosthetic valve infective endocarditis caused by staphylococcus to act on the biofilm. However, the use of this molecule is associated with numerous adverse effects (digestive disorders, hepatotoxicity, hypersensitivity…) and drug interactions, particularly common in patients with prosthetic valves. In a retrospective study comparing patients receiving antibiotic therapy with rifampin versus without rifampin in staphylococcal prosthetic infective endocarditis (Le Bot et al. CID 2021, PMID: 32706879), there was no difference in terms of mortality or relapse between the two groups, but a longer hospital length of stay in the rifampin-treated group.

The aim of this multicentre randomized controlled trial is to demonstrate the non-inferiority of a rifampin-free regimen compared to a rifampin-combined regimen.

ELIGIBILITY:
Inclusion Criteria:

* Definite infective endocarditis according to the 2023 Duke ISCVID criteria or confirmed by the endocarditis team if the endocarditis was classified as possible
* Prosthetic valve endocarditis
* At least one positive blood culture due to Staphylococcus sp (S. aureus or CoNS)
* After the first positive blood culture, at least one negative blood culture (after a minimum of 72 hours of incubation)
* Infective endocarditis due to Staphylococcus sp (S. aureus or coagulase negative staphylococci) susceptible to rifampin
* Antistaphylococcal treatment for endocarditis introduced less than 14 days ago. We do not consider all antibiotic received before the first positive blood culture
* Age ≥ 18-year-old
* Informed, written consent obtained from patient or from patient's near in kin
* Patient insured under a health insurance scheme
* Patient with adequate contraceptive measure

Exclusion Criteria:

* Presence of cardiovascular implanted electronic device with suspected device-related IE without removal of the device
* Expected duration of follow-up <6 months at the time of randomization
* Patient moribund (expected to die in next 48 hours with or without treatment)
* Patients already receiving more than 72 hours of rifampin for the endocarditis treatment prior to randomization
* Positive blood cultures less than 72 hours before randomization
* Medical history of infective endocarditis in the last 3 months
* True allergy to rifampin or a severe intolerance to rifampin
* Contraindication to rifampin
* Patients requiring treatment contraindicated or not recommended with rifampin or incompatible with the inducer effect of rifampicin according to the marketing authorisation.
* ALAT increase greater than 3 times the upper laboratory range
* Extreme weight (< 45 kg or > 150 kg)
* Patients with confirmed prosthetic vascular graft infection or orthopedic-device-related infection
* Patients treated with rifampin for infections other than endocarditis, such as tuberculosis
* Pregnancy or breastfeeding woman
* Inclusion in another drug clinical trial
* Patients who have already been included in the study for a previous episode of endocarditis
* Patients under court protection, guardianship or trusteeship
* Patients who do not speak or understand French language
* Patient unable to collect information in a daily journal
* Patient unable to understand a follow-up by phone contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate at 6 months | Up to 6 months
  Deaths of all causes from randomizaton until 6 months

SECONDARY OUTCOMES:
Microbiological failure | Up to 6 months
  Proportions of patients with at least one microbiological failure defined by bacteremia with the primary pathogen obtained during follow-up but before the end of curative treatment.
Relapse | Up to 12 months
  Proportions of patients with at least one relapse defined by bacteremia with the primary pathogen obtained during follow-up after the end of treatment of endocarditis until 6 months, then until 12 months.
Clinically evident embolic event | Up to 6 months
  Proportions of patients with at least one clinically evident embolic event (defined as secondary osteoarticular, splenic, brain or other symptomatic localizations) from randomization until 6 months.
Valvular surgery | Up to 12 months
  Proportions of patients with at least one valvular surgery at 6 months and at 12 months
Clinical failure | Up to 6 months
  Proportions of patients with clinical failure (defined by a composite criterion: all-cause mortality or microbiological failure or relapse or embolic event or valvular surgery) at 6 months.
Time to clinical failure | Up to 6 months
  Time between randomization and occurence of a clinical failure
Adverse events | Up to 6 months
  Proportions of patients with at least one adverse event grade III or IV related to treatment
Bleeding complications | Up to 6 months
  Proportions of patients with at least one bleeding complication
Lenght of stay in hospital | Up to 6 months
  Lenght of stay in hospital
Duration of curative antibiotic treatment for endocarditis | Up to 6 months
  Duration of curative antibiotic treatment for endocarditis
All-cause mortality rate at discharge, at 3 and at 12 months | Up to 12 months
  Deaths of all causes from randomization until discharge, then until 3 months and then until 12months
Readmission in hospitals | Up to 12 months
  Proportions of patients with at least one readmission in hospital (whatever the reason).
Reclassification of relapse or microbiological failure as reinfection. | Up to 12 months
  Proportions of patients with reclassification of relapse or microbiological failure as reinfection. To determine the proportion of relapses or microbiological failures that are in fact reinfections, the genome of the strain isolated at the time of the suspected microbiological failure or relapse will be compared with the genome of the strain isolated at the time of the initial infection. This will be performed by the national reference center for staphylococci based in Lyon CHU.
Cost-Effectiveness ratio | Up to 12 months
  Incremental cost-effectiveness ratio (cost per quality-adjusted life year (QALYs) gained)

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - CH metropole Savoie, Chambery, GHT Savoie-Belley, Site Aix les Bains, Aix-les-Bains
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Cardiologic hospital of Haut lévêque, Bordeaux
  - CHU Bordeaux, Haut Lévêque Hospital, Infectious disease department, Bordeaux
  - CHU Brest, Brest
  - AP-HP, Groupe hospitalier Henri Mondor, Créteil
  - CHU Dijon Bourgogne, Dijon
  - CHU Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHU Lyon, La Croix-Rousse Hospital, Infective disease department, Lyon
  - CHU Lyon, Louis Pradel Hospital, Cardiology Institute, Lyon
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Hôtel Dieu Hospital, Infective disease department, Nantes
  - CHU Nantes, Laennec Hospital, Cardiology department, Nantes
  - CHU Nice, Nice
  - CHR Orléans, Orléans
  - AP-HP hôpital St Antoine, Paris
  - AP-HP, Hôpital Pitié Salpétrière, Paris
  - AP-HP, hôpital Bichat-Claude Bernard, Paris
  - CH Pau, Pau
  - CHU Poitiers, Poitiers
  - CH intercommunal Cornouaille Quimper, Quimper
  - CHU Rennes, Rennes
  - CHU St-Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Purpan Hospital, Infectious disease department, Toulouse
  - CHU Toulouse, Rangueil Hospital, Cardiology department, Toulouse
  - CH Tourcoing, Tourcoing
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided